CLINICAL TRIAL: NCT01275547
Title: The Analgesic Effect of Combined Treatment With Intranasal S-Ketamine and Intranasal Midazolam Compared With Morphine Patient Controlled Analgesia in Spinal Surgery Patients
Brief Title: The Analgesic Effect of Combined Treatment With Intranasal S-ketamine and Intranasal Midazolam
Acronym: NASKEMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EKBB28/10
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Analgesia, Patient-controlled; Spinal Stenosis
Keywords: Patient controlled analgesia; Morphine; S-Ketamine intranasal; Midazolam intranasal
MeSH Terms: conditions — Agnosia; Spinal Stenosis | interventions — Esketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-ketamine & midazolam spray (Experimental): all 20 minutes as a patient controlled analgesia alternating s-ketamine / midazolam
  Interventions: Drug: s-ketamine & midazolam
- morphine, patient controlled analgesia (Active Comparator): morphine as an active comparator as a patient controlled analgesia system
  Interventions: Drug: Morphine PCA

INTERVENTIONS:
Drug: s-ketamine & midazolam — s-ketamine 6 mg intranasal midazolam 0.75 mg intranasal
  Arms: S-ketamine & midazolam spray
Drug: Morphine PCA — 2 mg Morphine i.v. all 12 minutes as a patient controlled system
  Arms: morphine, patient controlled analgesia

SUMMARY:
Introduction

Ketamine is an old and generally well accepted analgesic used in the intra- and perioperative setting. Several studies demonstrated the effectiveness of ketamine in the postoperative setting.

A new formulation of S-ketamine as an intranasal spray device was tested in our hospital in 8 healthy volunteers (unpublished data, EKBB 351/08). 20 mg of S-ketamine were administered intranasally and compared with S-ketamine i.v. and i.m.. None of the volunteers had serious adverse effects or complications. A preliminary data analysis shows a clear analgesic effect and good absorption of the intranasal S-ketamine.

As a next step we would like to investigate the effect of S-ketamine intranasal spray combined with midazolam intranasal spray in a group of postoperative spinal surgery patients. The rational for the combination of intranasal S-ketamine and midazolam is the well known midazolam antagonising effect of ketamine induced psychomimetic adverse effects. Furthermore we know from other studies (EKBB 106/06) that midazolam intranasal spray has relaxant and anxiolytic effects. As far as we know, this is the first study which will examine the combination of S-ketamine and midazolam intranasal sprays in adult patients.

Study work plan

This prospective, randomized, double-blinded non inferiority study will address pain ratings and patient satisfaction in a postoperative setting in two treatment scenarios:

1. Alternating S-ketamine intranasal unit-dose spray (6 mg per dose) with midazolam intranasal spray (0.75 mg per dose) patient controlled application with a lock-out interval of 20 minutes between two applications and placebo patient controlled analgesia (PCA) with a lock-out interval of 12 minutes with saline 0.9% i.v. for 72 hours or until 40 unit-dose sprays are delivered
2. PCA with 2 mg morphine with a lock-out interval of 12 minutes i.v. with placebo intranasal spray (saline 0.9% + chitosan) with a minimum lock-out interval of 20 minutes for 72 hours or until 40 unit-dose sprays are delivered

Patient number

We will examine 36 patients, 18 patients in each group. The study duration for an individual patient will be at latest 72 hours, the total study duration is 4 to 5 months.

Study importance

An intranasal spray is an ideal application form for surgery patients, either in- or outpatients. On the other hand, ketamine and S-ketamine is quite often used in the perioperative setting as a rescue analgesic. In higher doses it could be used as an emergency tool in emergency prehospital medicine. In the perioperative setting it is important to evaluate the efficacy and safety of S-ketamine intranasal spray combined with midazolam intranasal spray in patients.

If our study shows that S-ketamine intranasal spray is effective as an analgesic and has good patient acceptance, S-ketamine intranasal spay could be considered as an alternative, completely non-invasive analgesic procedure in a postoperative outpatient setting. As a consequence development of a nasal multidose-applicator combining S-ketamine and midazolam would be of interest.

ELIGIBILITY:
Inclusion Criteria:

* Spinal surgery patients with:

  * decompression because of spinal stenosis
  * laminectomy because of spinal stenosis
* Age > 18 years
* BMI 18 - 39.9 (kg/m2)

Exclusion Criteria:

* Patients unable to give written informed consent

  * Known drug allergies or intolerance to the study medications morphine, midazolam, ketamine, paracetamol or metamizol
  * Known allergy to crustacea or chitosan
  * Patients using snuff at a regularly basis
  * Recreational drug addiction or abuse
  * Preexisting opioid (tramadol excluded), ketamine or midazolam therapy
  * General physical condition ≥ ASA IV
  * Serious intranasal or epipharyngeal problems
  * Mental / psychiatric disorder
  * Pregnancy
  * Patients with renal failure (clearance < 30 ml/min)
  * Patients with liver failure (MELD score > 25) Investigational Product Morphine / S-ketamine / midazolam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale 24 hours after surgery | 24 hours
  NRS after 24 hours after finishing surgery

SECONDARY OUTCOMES:
Amount of PCA boli | 72 hours
  Amount of demanded / delivered unit doses of intranasal S-ketamine
  / midazolam or morphine PCA-boli

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland, Basel, Canton of Basel-City, Switzerland